CLINICAL TRIAL: NCT04031716
Title: Genetic, Epigenetic, Psychosocial, and Biological Determinants of Post-surgical Pain After Pectus or Spine Surgery
Brief Title: Comprehensive Study of Post-surgical Pain After Pectus or Spine Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-5817
Record Dates: First submitted 2018-09-20; First posted 2019-07-24 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pain, Postoperative; Excavatum, Pectus; Scoliosis Idiopathic
Keywords: Meditation; Pectus Excavatum; Scoliosis
MeSH Terms: conditions — Pain, Postoperative; Funnel Chest; Scoliosis | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: All participants will receive standard perioperative care, anesthetic management, and postoperative pain management per institutional standardized practices. Participants will be randomized into either the Meditation or Control Groups, as deemed appropriate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Participants in the control group will receive present standard of care, which includes an assessment of participant/family needs by integrative care after surgery, as well as standard holistic health care by a licensed/certified holistic health specialist. They will not receive the MUSETM focused-attention meditation training or intervention protocol.
- Meditation (Experimental): Participants randomized to receive focused-attention meditation training will attend a preoperative training session, provided by a licensed/certified Holistic Health Specialist. The content will include an age appropriate explanation of focused-attention meditation, using breath as the focus; set-up and utilization of the MUSETM headband; and experiential practices. The goal of the intervention is to increase mindfulness (i.e., moment-to-moment, non-judgmental and non-reactive awareness of sensations, emotions, and thoughts), provide self-regulation strategies, and promote healthy and adaptive responses to stress.
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — Participants assigned to the Meditation intervention will receive focused attention meditation training preoperatively, and encouraged to meditate for 20 minutes per day before surgery. In the postoperative inpatient period, the participants will be offered standard holistic health care, reinforcement of meditation training, and encouragement to practice at least 20 minutes of guided focused-attention meditation with breath as their focus, utilizing the MUSETM headband for bio-feedback, every day during their hospital stay. They will be asked to continue using the MUSETM neurofeedback-assisted meditation after hospital discharge, until their visit to repeat pain testing, at which time they will return the MUSETM headband.
  Arms: Meditation

SUMMARY:
This will be a prospective study to determine the association between specific genotypes, epigenetics, behavioral, social and biological factors, with the phenotypes, defined by pain perception, postoperative pain, analgesic effects, side effects to perioperative analgesics, chronic postoperative pain, and gene expression in patients following pectus excavatum repair.

DETAILED DESCRIPTION:
This study will be a clinical prospective study. It is observational for all aims except with regard to the Meditation Intervention, which will be limited to 100 pectus and 100 spine participants (randomized to 50/50 in each arm). We will recruit 600 qualifying participants over the study period to acquire the necessary data to derive a predictive model matching phenotype to genotype. This study will not interfere with the standard anesthetic or perioperative care except for blood sampling from an indwelling line, and the use of additional integrative health procedures (focused-attention meditation guidance, as well as routine massage and breathing techniques) for the randomized meditation group. Research staff will administer psychosocial and somatosensory assessments, as well as record relevant data from participant's medical records. Integrative health will assist in teaching focused-attention meditation to the randomized meditation participants in the preoperative phase. Actigraphy devices will be provided to all participants, and MUSETM to those in the randomized meditation group. The pain team, in accordance with the Pectus Pain Management Protocol, will direct perioperative pain management.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 years of age through adulthood
* Diagnosis of pectus excavatum or adolescent idiopathic scoliosis
* Scheduled for endoscopic pectus excavatum repair or spine fusion

Exclusion Criteria:

* History of or active renal or liver disease
* Major surgery requiring opioids in the last 5 years
* Severe respiratory problems (such as obstructive sleep apnea, cystic fibrosis, pulmonary fibrosis, or pneumonia within the last month)
* Cardiac conditions including, but not limited to, cyanotic heart disease, hypoplastic left ventricle, arrhythmia, hypertension with ongoing treatment, Kawasaki disease, or cardiomyopathies. Participants with asymptomatic valvular lesions or defects may be included
* History of seizures currently treated on medication (participants off medication and seizure free for greater than one year may be included)
* Taking no more than two concomitant medications known to induce or inhibit CYP2D6 activity, including paroxetine, fluoxetine, cimetidine, and duloxetine
* Needing postoperative ventilation or intraoperative cardiac bypass standby
* BMI >35
* Pregnant or breastfeeding females
* Non-English speaking
* Definite developmental delay

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-07-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score trajectory | 1 year
  Pain scores will be collected preoperatively through 1 year postoperatively
Changes in self-reported psychosocial scores (including anxiety, pain, coping, physical limitation, etc.) | 1 year
  Psychosocial measures will be collected preoperatively through 1 year postoperatively
Changes in heart rate variability | 8 weeks
  Heart rate variability will be assessed preoperatively and postoperatively
Changes in mean amplitude values for lower, upper, and entire alpha frequency bands by group (intervention/no intervention) and time (pre-surgery/post-surgery) | 8 weeks
  Brain activity will be assessed preoperatively and postoperatively
Changes in evoked response potentials (ERPs) during meditation and experimental pain tasks | 8 weeks
  Brain activity will be assessed preoperatively and postoperatively
Changes in sleep efficiency/duration (actigraphy) and self-reported sleep quality | 8 weeks
  Sleep efficiency and quality will be assessed preoperatively and postoperatively
Incidence of side-effect measures | 72 hours postoperatively
  Incidences of respiratory depression, sedation, postoperative nausea and vomiting will be collected during the recovery phase

SECONDARY OUTCOMES:
Changes in pressure pain threshold, conditioned pain modulation, tactile discrimination, and temporal summation index | 8 weeks
  Quantitative sensory testing will be assessed preoperatively and postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Chidambaran, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with additional internal or external data warehouses/investigators. These include but are not limited to the i2b2-Research Data Warehouse protocol at CCHMC (IRB 2008-0834) for the purpose of linking this data to de-identified copies of the participants' electronic medical records via an i2b2 database. The resulting de-identified i2b2 database will not be part of this research, and will be used to explore secondary phenotypes in future research studies and the NIH-db-GaP (Database of Genotypes and Phenotypes).

REFERENCES:
- [Background] Perquin CW, Hazebroek-Kampschreur AAJM, Hunfeld JAM, Bohnen AM, van Suijlekom-Smit LWA, Passchier J, van der Wouden JC. Pain in children and adolescents: a common experience. Pain. 2000 Jul;87(1):51-58. doi: 10.1016/S0304-3959(00)00269-4. PMID 10863045
- [Background] Duedahl TH, Hansen EH. A qualitative systematic review of morphine treatment in children with postoperative pain. Paediatr Anaesth. 2007 Aug;17(8):756-74. doi: 10.1111/j.1460-9592.2007.02213.x. PMID 17596221
- [Background] Beaulieu P, Cyrenne L, Mathews S, Villeneuve E, Vischoff D. Patient-controlled analgesia after spinal fusion for idiopathic scoliosis. Int Orthop. 1996;20(5):295-9. doi: 10.1007/s002640050081. PMID 8930721
- [Background] Klepstad P, Dale O, Skorpen F, Borchgrevink PC, Kaasa S. Genetic variability and clinical efficacy of morphine. Acta Anaesthesiol Scand. 2005 Aug;49(7):902-8. doi: 10.1111/j.1399-6576.2005.00772.x. PMID 16045647
- [Background] Berde CB, Sethna NF. Analgesics for the treatment of pain in children. N Engl J Med. 2002 Oct 3;347(14):1094-103. doi: 10.1056/NEJMra012626. No abstract available. PMID 12362012
- [Background] Kotzer AM, Foster R. Children's use of PCA following spinal fusion. Orthop Nurs. 2000 Sep-Oct;19(5):19-27; quiz 28-30. doi: 10.1097/00006416-200019050-00005. PMID 11153382
- [Background] Macrae WA, Davies HTO. Chronic postsurgical pain. In: Crombie IK, editor. Epidemiology of Pain. Seattle: IASP Press, 1999; p. 125-142.
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Macrae WA. Chronic post-surgical pain: 10 years on. Br J Anaesth. 2008 Jul;101(1):77-86. doi: 10.1093/bja/aen099. Epub 2008 Apr 22. PMID 18434337
- [Background] Gaskin DJ, Richard P. The economic costs of pain in the United States. J Pain. 2012 Aug;13(8):715-24. doi: 10.1016/j.jpain.2012.03.009. Epub 2012 May 16. PMID 22607834
- [Background] Page MG, Stinson J, Campbell F, Isaac L, Katz J. Identification of pain-related psychological risk factors for the development and maintenance of pediatric chronic postsurgical pain. J Pain Res. 2013;6:167-80. doi: 10.2147/JPR.S40846. Epub 2013 Mar 5. PMID 23503375
- [Background] Nakanii M, Nanba T, Uemura S. Pain Caused by the Pectus Bar Implant after the Nuss Procedure for Pectus Excavatum among Junior High and High School Children. Kawasaki Journal of Medical Welfare 2011; 17(1): 15-21.
- [Background] Uemura S CY. Nuss Procedure for Pectus Excavatum and the Operative Results. Pedia Surg 2003; 35(6): 665-71.
- [Background] Hocking LJ; Generation Scotland; Morris AD, Dominiczak AF, Porteous DJ, Smith BH. Heritability of chronic pain in 2195 extended families. Eur J Pain. 2012 Aug;16(7):1053-63. doi: 10.1002/j.1532-2149.2011.00095.x. Epub 2012 Jan 26. PMID 22337623
- [Background] Connelly M, Fulmer RD, Prohaska J, Anson L, Dryer L, Thomas V, Ariagno JE, Price N, Schwend R. Predictors of postoperative pain trajectories in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2014 Feb 1;39(3):E174-81. doi: 10.1097/BRS.0000000000000099. PMID 24173016
- [Background] Rabbitts JA, Zhou C, Groenewald CB, Durkin L, Palermo TM. Trajectories of postsurgical pain in children: risk factors and impact of late pain recovery on long-term health outcomes after major surgery. Pain. 2015 Nov;156(11):2383-2389. doi: 10.1097/j.pain.0000000000000281. PMID 26381701
- [Background] Rabbitts JA, Groenewald CB, Tai GG, Palermo TM. Presurgical psychosocial predictors of acute postsurgical pain and quality of life in children undergoing major surgery. J Pain. 2015 Mar;16(3):226-34. doi: 10.1016/j.jpain.2014.11.015. Epub 2014 Dec 22. PMID 25540939
- [Background] Page MG, Campbell F, Isaac L, Stinson J, Katz J. Parental risk factors for the development of pediatric acute and chronic postsurgical pain: a longitudinal study. J Pain Res. 2013 Sep 30;6:727-41. doi: 10.2147/JPR.S51055. eCollection 2013. PMID 24109194
- [Background] Guite JW, McCue RL, Sherker JL, Sherry DD, Rose JB. Relationships among pain, protective parental responses, and disability for adolescents with chronic musculoskeletal pain: the mediating role of pain catastrophizing. Clin J Pain. 2011 Nov-Dec;27(9):775-81. doi: 10.1097/AJP.0b013e31821d8fb4. PMID 21593664
- [Background] Rakvag TT, Klepstad P, Baar C, Kvam TM, Dale O, Kaasa S, Krokan HE, Skorpen F. The Val158Met polymorphism of the human catechol-O-methyltransferase (COMT) gene may influence morphine requirements in cancer pain patients. Pain. 2005 Jul;116(1-2):73-8. doi: 10.1016/j.pain.2005.03.032. PMID 15927391
- [Background] Nackley AG, Tan KS, Fecho K, Flood P, Diatchenko L, Maixner W. Catechol-O-methyltransferase inhibition increases pain sensitivity through activation of both beta2- and beta3-adrenergic receptors. Pain. 2007 Apr;128(3):199-208. doi: 10.1016/j.pain.2006.09.022. Epub 2006 Nov 7. PMID 17084978
- [Background] Diatchenko L, Nackley AG, Slade GD, Bhalang K, Belfer I, Max MB, Goldman D, Maixner W. Catechol-O-methyltransferase gene polymorphisms are associated with multiple pain-evoking stimuli. Pain. 2006 Dec 5;125(3):216-224. doi: 10.1016/j.pain.2006.05.024. Epub 2006 Jul 11. PMID 16837133
- [Background] Diatchenko L, Slade GD, Nackley AG, Bhalang K, Sigurdsson A, Belfer I, Goldman D, Xu K, Shabalina SA, Shagin D, Max MB, Makarov SS, Maixner W. Genetic basis for individual variations in pain perception and the development of a chronic pain condition. Hum Mol Genet. 2005 Jan 1;14(1):135-43. doi: 10.1093/hmg/ddi013. Epub 2004 Nov 10. PMID 15537663
- [Background] Zubieta JK, Heitzeg MM, Smith YR, Bueller JA, Xu K, Xu Y, Koeppe RA, Stohler CS, Goldman D. COMT val158met genotype affects mu-opioid neurotransmitter responses to a pain stressor. Science. 2003 Feb 21;299(5610):1240-3. doi: 10.1126/science.1078546. PMID 12595695
- [Background] Oertel BG, Schmidt R, Schneider A, Geisslinger G, Lotsch J. The mu-opioid receptor gene polymorphism 118A>G depletes alfentanil-induced analgesia and protects against respiratory depression in homozygous carriers. Pharmacogenet Genomics. 2006 Sep;16(9):625-36. doi: 10.1097/01.fpc.0000220566.90466.a2. PMID 16906017
- [Background] Chou WY, Wang CH, Liu PH, Liu CC, Tseng CC, Jawan B. Human opioid receptor A118G polymorphism affects intravenous patient-controlled analgesia morphine consumption after total abdominal hysterectomy. Anesthesiology. 2006 Aug;105(2):334-7. doi: 10.1097/00000542-200608000-00016. PMID 16871067
- [Background] Chou WY, Yang LC, Lu HF, Ko JY, Wang CH, Lin SH, Lee TH, Concejero A, Hsu CJ. Association of mu-opioid receptor gene polymorphism (A118G) with variations in morphine consumption for analgesia after total knee arthroplasty. Acta Anaesthesiol Scand. 2006 Aug;50(7):787-92. doi: 10.1111/j.1399-6576.2006.01058.x. PMID 16879459
- [Background] Klepstad P, Rakvag TT, Kaasa S, Holthe M, Dale O, Borchgrevink PC, Baar C, Vikan T, Krokan HE, Skorpen F. The 118 A > G polymorphism in the human mu-opioid receptor gene may increase morphine requirements in patients with pain caused by malignant disease. Acta Anaesthesiol Scand. 2004 Nov;48(10):1232-9. doi: 10.1111/j.1399-6576.2004.00517.x. PMID 15504181
- [Background] Reyes-Gibby CC, Shete S, Rakvag T, Bhat SV, Skorpen F, Bruera E, Kaasa S, Klepstad P. Exploring joint effects of genes and the clinical efficacy of morphine for cancer pain: OPRM1 and COMT gene. Pain. 2007 Jul;130(1-2):25-30. doi: 10.1016/j.pain.2006.10.023. Epub 2006 Dec 6. PMID 17156920
- [Background] Pasternak GW. The pharmacology of mu analgesics: from patients to genes. Neuroscientist. 2001 Jun;7(3):220-31. doi: 10.1177/107385840100700307. PMID 11499401
- [Background] Coulbault L, Beaussier M, Verstuyft C, Weickmans H, Dubert L, Tregouet D, Descot C, Parc Y, Lienhart A, Jaillon P, Becquemont L. Environmental and genetic factors associated with morphine response in the postoperative period. Clin Pharmacol Ther. 2006 Apr;79(4):316-24. doi: 10.1016/j.clpt.2006.01.007. PMID 16580900
- [Background] Coller JK, Barratt DT, Dahlen K, Loennechen MH, Somogyi AA. ABCB1 genetic variability and methadone dosage requirements in opioid-dependent individuals. Clin Pharmacol Ther. 2006 Dec;80(6):682-90. doi: 10.1016/j.clpt.2006.09.011. PMID 17178268
- [Background] Hemmings SM, Martin LI, Klopper M, van der Merwe L, Aitken L, de Wit E, Black GF, Hoal EG, Walzl G, Seedat S. BDNF Val66Met and DRD2 Taq1A polymorphisms interact to influence PTSD symptom severity: a preliminary investigation in a South African population. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Jan 10;40:273-80. doi: 10.1016/j.pnpbp.2012.10.011. Epub 2012 Oct 26. PMID 23103549
- [Background] Kukreti R, Tripathi S, Bhatnagar P, Gupta S, Chauhan C, Kubendran S, Janardhan Reddy YC, Jain S, Brahmachari SK. Association of DRD2 gene variant with schizophrenia. Neurosci Lett. 2006 Jan 9;392(1-2):68-71. doi: 10.1016/j.neulet.2005.08.059. Epub 2005 Sep 23. PMID 16183199
- [Background] Barratt DT, Coller JK, Somogyi AA. Association between the DRD2 A1 allele and response to methadone and buprenorphine maintenance treatments. Am J Med Genet B Neuropsychiatr Genet. 2006 Jun 5;141B(4):323-31. doi: 10.1002/ajmg.b.30319. PMID 16583408
- [Background] Lawford BR, Young R, Noble EP, Kann B, Ritchie T. The D2 dopamine receptor (DRD2) gene is associated with co-morbid depression, anxiety and social dysfunction in untreated veterans with post-traumatic stress disorder. Eur Psychiatry. 2006 Apr;21(3):180-5. doi: 10.1016/j.eurpsy.2005.01.006. PMID 16632165
- [Background] George SZ, Wallace MR, Wright TW, Moser MW, Greenfield WH 3rd, Sack BK, Herbstman DM, Fillingim RB. Evidence for a biopsychosocial influence on shoulder pain: pain catastrophizing and catechol-O-methyltransferase (COMT) diplotype predict clinical pain ratings. Pain. 2008 May;136(1-2):53-61. doi: 10.1016/j.pain.2007.06.019. Epub 2007 Aug 7. PMID 17686583
- [Background] Belfer I, Dai F, Kehlet H, Finelli P, Qin L, Bittner R, Aasvang EK. Association of functional variations in COMT and GCH1 genes with postherniotomy pain and related impairment. Pain. 2015 Feb;156(2):273-279. doi: 10.1097/01.j.pain.0000460307.48701.b0. PMID 25599448
- [Background] Diatchenko L, Anderson AD, Slade GD, Fillingim RB, Shabalina SA, Higgins TJ, Sama S, Belfer I, Goldman D, Max MB, Weir BS, Maixner W. Three major haplotypes of the beta2 adrenergic receptor define psychological profile, blood pressure, and the risk for development of a common musculoskeletal pain disorder. Am J Med Genet B Neuropsychiatr Genet. 2006 Jul 5;141B(5):449-62. doi: 10.1002/ajmg.b.30324. PMID 16741943
- [Background] Gordon JA, Hen R. Genetic approaches to the study of anxiety. Annu Rev Neurosci. 2004;27:193-222. doi: 10.1146/annurev.neuro.27.070203.144212. PMID 15217331
- [Background] Kolesnikov Y, Gabovits B, Levin A, Veske A, Qin L, Dai F, Belfer I. Chronic pain after lower abdominal surgery: do catechol-O-methyl transferase/opioid receptor mu-1 polymorphisms contribute? Mol Pain. 2013 Apr 8;9:19. doi: 10.1186/1744-8069-9-19. PMID 23566343
- [Background] Tegeder I, Costigan M, Griffin RS, Abele A, Belfer I, Schmidt H, Ehnert C, Nejim J, Marian C, Scholz J, Wu T, Allchorne A, Diatchenko L, Binshtok AM, Goldman D, Adolph J, Sama S, Atlas SJ, Carlezon WA, Parsegian A, Lotsch J, Fillingim RB, Maixner W, Geisslinger G, Max MB, Woolf CJ. GTP cyclohydrolase and tetrahydrobiopterin regulate pain sensitivity and persistence. Nat Med. 2006 Nov;12(11):1269-77. doi: 10.1038/nm1490. Epub 2006 Oct 22. PMID 17057711
- [Background] Jayamanne A, Greenwood R, Mitchell VA, Aslan S, Piomelli D, Vaughan CW. Actions of the FAAH inhibitor URB597 in neuropathic and inflammatory chronic pain models. Br J Pharmacol. 2006 Feb;147(3):281-8. doi: 10.1038/sj.bjp.0706510. PMID 16331291
- [Background] Sia AT, Sng BL, Lim EC, Law H, Tan EC. The influence of ATP-binding cassette sub-family B member -1 (ABCB1) genetic polymorphisms on acute and chronic pain after intrathecal morphine for caesarean section: a prospective cohort study. Int J Obstet Anesth. 2010 Jul;19(3):254-60. doi: 10.1016/j.ijoa.2010.03.001. Epub 2010 Jun 2. PMID 20627697
- [Background] Noponen-Hietala N, Virtanen I, Karttunen R, Schwenke S, Jakkula E, Li H, Merikivi R, Barral S, Ott J, Karppinen J, Ala-Kokko L. Genetic variations in IL6 associate with intervertebral disc disease characterized by sciatica. Pain. 2005 Mar;114(1-2):186-94. doi: 10.1016/j.pain.2004.12.015. Epub 2005 Jan 22. PMID 15733644
- [Background] George SZ, Parr JJ, Wallace MR, Wu SS, Borsa PA, Dai Y, Fillingim RB. Inflammatory genes and psychological factors predict induced shoulder pain phenotype. Med Sci Sports Exerc. 2014 Oct;46(10):1871-81. doi: 10.1249/MSS.0000000000000328. PMID 24598699
- [Background] Banik RK, Brennan TJ. Trpv1 mediates spontaneous firing and heat sensitization of cutaneous primary afferents after plantar incision. Pain. 2009 Jan;141(1-2):41-51. doi: 10.1016/j.pain.2008.10.004. Epub 2008 Nov 17. PMID 19010598
- [Background] Reimann F, Cox JJ, Belfer I, Diatchenko L, Zaykin DV, McHale DP, Drenth JP, Dai F, Wheeler J, Sanders F, Wood L, Wu TX, Karppinen J, Nikolajsen L, Mannikko M, Max MB, Kiselycznyk C, Poddar M, Te Morsche RH, Smith S, Gibson D, Kelempisioti A, Maixner W, Gribble FM, Woods CG. Pain perception is altered by a nucleotide polymorphism in SCN9A. Proc Natl Acad Sci U S A. 2010 Mar 16;107(11):5148-53. doi: 10.1073/pnas.0913181107. Epub 2010 Mar 8. PMID 20212137
- [Background] Young EE, Lariviere WR, Belfer I. Genetic basis of pain variability: recent advances. J Med Genet. 2012 Jan;49(1):1-9. doi: 10.1136/jmedgenet-2011-100386. Epub 2011 Nov 5. PMID 22058430
- [Background] Crow M, Denk F, McMahon SB. Genes and epigenetic processes as prospective pain targets. Genome Med. 2013 Feb 15;5(2):12. doi: 10.1186/gm416. eCollection 2013. PMID 23409739
- [Background] Hwang CK, Song KY, Kim CS, Choi HS, Guo XH, Law PY, Wei LN, Loh HH. Evidence of endogenous mu opioid receptor regulation by epigenetic control of the promoters. Mol Cell Biol. 2007 Jul;27(13):4720-36. doi: 10.1128/MCB.00073-07. Epub 2007 Apr 23. PMID 17452465
- [Background] Angst MS, Phillips NG, Drover DR, Tingle M, Ray A, Swan GE, Lazzeroni LC, Clark DJ. Pain sensitivity and opioid analgesia: a pharmacogenomic twin study. Pain. 2012 Jul;153(7):1397-1409. doi: 10.1016/j.pain.2012.02.022. Epub 2012 Mar 22. PMID 22444188
- [Background] Norbury TA, MacGregor AJ, Urwin J, Spector TD, McMahon SB. Heritability of responses to painful stimuli in women: a classical twin study. Brain. 2007 Nov;130(Pt 11):3041-9. doi: 10.1093/brain/awm233. Epub 2007 Oct 11. PMID 17932101
- [Background] Graff J, Kim D, Dobbin MM, Tsai LH. Epigenetic regulation of gene expression in physiological and pathological brain processes. Physiol Rev. 2011 Apr;91(2):603-49. doi: 10.1152/physrev.00012.2010. PMID 21527733
- [Background] Vucetic Z, Kimmel J, Reyes TM. Chronic high-fat diet drives postnatal epigenetic regulation of mu-opioid receptor in the brain. Neuropsychopharmacology. 2011 May;36(6):1199-206. doi: 10.1038/npp.2011.4. Epub 2011 Feb 16. PMID 21326195
- [Background] Buchheit T, Van de Ven T, Shaw A. Epigenetics and the transition from acute to chronic pain. Pain Med. 2012 Nov;13(11):1474-90. doi: 10.1111/j.1526-4637.2012.01488.x. Epub 2012 Sep 14. PMID 22978429
- [Background] Hoofwijk DM, van Reij RR, Rutten BP, Kenis G, Buhre WF, Joosten EA. Genetic polymorphisms and their association with the prevalence and severity of chronic postsurgical pain: a systematic review. Br J Anaesth. 2016 Dec;117(6):708-719. doi: 10.1093/bja/aew378. PMID 27956669
- [Background] Montes A, Roca G, Sabate S, Lao JI, Navarro A, Cantillo J, Canet J; GENDOLCAT Study Group. Genetic and Clinical Factors Associated with Chronic Postsurgical Pain after Hernia Repair, Hysterectomy, and Thoracotomy: A Two-year Multicenter Cohort Study. Anesthesiology. 2015 May;122(5):1123-41. doi: 10.1097/ALN.0000000000000611. PMID 25985024
- [Background] Katz J, Seltzer Z. Transition from acute to chronic postsurgical pain: risk factors and protective factors. Expert Rev Neurother. 2009 May;9(5):723-44. doi: 10.1586/ern.09.20. PMID 19402781
- [Background] Oertel B, Lotsch J. Genetic mutations that prevent pain: implications for future pain medication. Pharmacogenomics. 2008 Feb;9(2):179-94. doi: 10.2217/14622416.9.2.179. PMID 18370847
- [Background] Ushijima T, Nakajima T, Maekita T. DNA methylation as a marker for the past and future. J Gastroenterol. 2006 May;41(5):401-7. doi: 10.1007/s00535-006-1846-6. PMID 16799880
- [Background] Denk F, McMahon SB. Chronic pain: emerging evidence for the involvement of epigenetics. Neuron. 2012 Feb 9;73(3):435-44. doi: 10.1016/j.neuron.2012.01.012. PMID 22325197
- [Background] Oertel BG, Doehring A, Roskam B, Kettner M, Hackmann N, Ferreiros N, Schmidt PH, Lotsch J. Genetic-epigenetic interaction modulates mu-opioid receptor regulation. Hum Mol Genet. 2012 Nov 1;21(21):4751-60. doi: 10.1093/hmg/dds314. Epub 2012 Aug 8. PMID 22875838
- [Background] Chorbov VM, Todorov AA, Lynskey MT, Cicero TJ. Elevated levels of DNA methylation at the OPRM1 promoter in blood and sperm from male opioid addicts. J Opioid Manag. 2011 Jul-Aug;7(4):258-64. doi: 10.5055/jom.2011.0067. PMID 21957825
- [Background] Nielsen DA, Yuferov V, Hamon S, Jackson C, Ho A, Ott J, Kreek MJ. Increased OPRM1 DNA methylation in lymphocytes of methadone-maintained former heroin addicts. Neuropsychopharmacology. 2009 Mar;34(4):867-73. doi: 10.1038/npp.2008.108. Epub 2008 Jul 23. PMID 18650805
- [Background] Davies MN, Volta M, Pidsley R, Lunnon K, Dixit A, Lovestone S, Coarfa C, Harris RA, Milosavljevic A, Troakes C, Al-Sarraj S, Dobson R, Schalkwyk LC, Mill J. Functional annotation of the human brain methylome identifies tissue-specific epigenetic variation across brain and blood. Genome Biol. 2012 Jun 15;13(6):R43. doi: 10.1186/gb-2012-13-6-r43. PMID 22703893
- [Background] Roth TL. Epigenetic mechanisms in the development of behavior: advances, challenges, and future promises of a new field. Dev Psychopathol. 2013 Nov;25(4 Pt 2):1279-91. doi: 10.1017/S0954579413000618. PMID 24342840
- [Background] Chen ZX, Riggs AD. DNA methylation and demethylation in mammals. J Biol Chem. 2011 May 27;286(21):18347-53. doi: 10.1074/jbc.R110.205286. Epub 2011 Mar 24. PMID 21454628
- [Background] Orphanides G, Reinberg D. A unified theory of gene expression. Cell. 2002 Feb 22;108(4):439-51. doi: 10.1016/s0092-8674(02)00655-4. PMID 11909516
- [Background] Bird A. Perceptions of epigenetics. Nature. 2007 May 24;447(7143):396-8. doi: 10.1038/nature05913. PMID 17522671
- [Background] Ueda H, Uchida H. Epigenetic modification in neuropathic pain. Curr Pharm Des. 2015;21(7):849-67. doi: 10.2174/1381612820666141027113923. PMID 25345610
- [Background] Uchida H, Matsushita Y, Ueda H. Epigenetic regulation of BDNF expression in the primary sensory neurons after peripheral nerve injury: implications in the development of neuropathic pain. Neuroscience. 2013 Jun 14;240:147-54. doi: 10.1016/j.neuroscience.2013.02.053. Epub 2013 Mar 4. PMID 23466809
- [Background] Uchida H, Ma L, Ueda H. Epigenetic gene silencing underlies C-fiber dysfunctions in neuropathic pain. J Neurosci. 2010 Mar 31;30(13):4806-14. doi: 10.1523/JNEUROSCI.5541-09.2010. PMID 20357131
- [Background] Lotsch J, Oertel BG, Ultsch A. Human models of pain for the prediction of clinical analgesia. Pain. 2014 Oct;155(10):2014-21. doi: 10.1016/j.pain.2014.07.003. Epub 2014 Jul 11. PMID 25020003
- [Background] Blankenburg M, Boekens H, Hechler T, Maier C, Krumova E, Scherens A, Magerl W, Aksu F, Zernikow B. Reference values for quantitative sensory testing in children and adolescents: developmental and gender differences of somatosensory perception. Pain. 2010 Apr;149(1):76-88. doi: 10.1016/j.pain.2010.01.011. Epub 2010 Feb 6. PMID 20138430
- [Background] Hirschfeld G, Zernikow B, Kraemer N, Hechler T, Aksu F, Krumova E, Maier C, Magerl W, Blankenburg M. Development of somatosensory perception in children: a longitudinal QST-study. Neuropediatrics. 2012 Feb;43(1):10-6. doi: 10.1055/s-0032-1307450. Epub 2012 Mar 19. PMID 22430155
- [Background] Birnie KA, Caes L, Wilson AC, Williams SE, Chambers CT. A practical guide and perspectives on the use of experimental pain modalities with children and adolescents. Pain Manag. 2014 Mar;4(2):97-111. doi: 10.2217/pmt.13.72. PMID 24641434
- [Background] Chu LF, Clark DJ, Angst MS. Opioid tolerance and hyperalgesia in chronic pain patients after one month of oral morphine therapy: a preliminary prospective study. J Pain. 2006 Jan;7(1):43-8. doi: 10.1016/j.jpain.2005.08.001. PMID 16414554
- [Background] Petersen KK, Arendt-Nielsen L, Simonsen O, Wilder-Smith O, Laursen MB. Presurgical assessment of temporal summation of pain predicts the development of chronic postoperative pain 12 months after total knee replacement. Pain. 2015 Jan;156(1):55-61. doi: 10.1016/j.pain.0000000000000022. PMID 25599301
- [Background] Weissman-Fogel I, Granovsky Y, Crispel Y, Ben-Nun A, Best LA, Yarnitsky D, Granot M. Enhanced presurgical pain temporal summation response predicts post-thoracotomy pain intensity during the acute postoperative phase. J Pain. 2009 Jun;10(6):628-36. doi: 10.1016/j.jpain.2008.12.009. Epub 2009 Apr 23. PMID 19398382
- [Background] Rabbitts JA, Zhou C, Narayanan A, Palermo TM. Longitudinal and Temporal Associations Between Daily Pain and Sleep Patterns After Major Pediatric Surgery. J Pain. 2017 Jun;18(6):656-663. doi: 10.1016/j.jpain.2017.01.004. Epub 2017 Jan 26. PMID 28131699
- [Background] Kanstrup M, Holmstrom L, Ringstrom R, Wicksell RK. Insomnia in paediatric chronic pain and its impact on depression and functional disability. Eur J Pain. 2014 Sep;18(8):1094-102. doi: 10.1002/j.1532-2149.2013.00450.x. Epub 2014 Jan 20. PMID 24443275
- [Background] Chung KF, Kan KK, Yeung WF. Assessing insomnia in adolescents: comparison of Insomnia Severity Index, Athens Insomnia Scale and Sleep Quality Index. Sleep Med. 2011 May;12(5):463-70. doi: 10.1016/j.sleep.2010.09.019. Epub 2011 Apr 13. PMID 21493134
- [Background] Berntson GG, Bigger JT Jr, Eckberg DL, Grossman P, Kaufmann PG, Malik M, Nagaraja HN, Porges SW, Saul JP, Stone PH, van der Molen MW. Heart rate variability: origins, methods, and interpretive caveats. Psychophysiology. 1997 Nov;34(6):623-48. doi: 10.1111/j.1469-8986.1997.tb02140.x. PMID 9401419
- [Background] Katahira K, Fujimura T, Matsuda YT, Okanoya K, Okada M. Individual differences in heart rate variability are associated with the avoidance of negative emotional events. Biol Psychol. 2014 Dec;103:322-31. doi: 10.1016/j.biopsycho.2014.10.007. Epub 2014 Oct 18. PMID 25457639
- [Background] Danev S, Radneva R, Zlatarov I. Changes in heart rate variability due to informational, physical and emotional load, in laboratory and field conditions. Act Nerv Super (Praha). 1975 Sep;17(3):187-8. No abstract available. PMID 1199687
- [Background] Nahman-Averbuch H, Coghill RC. Pain-autonomic relationships: implications for experimental design and the search for an "objective marker" for pain. Pain. 2017 Nov;158(11):2064-2065. doi: 10.1097/j.pain.0000000000001035. No abstract available. PMID 28858987
- [Background] Nahman-Averbuch H, Sprecher E, Jacob G, Yarnitsky D. The Relationships Between Parasympathetic Function and Pain Perception: The Role of Anxiety. Pain Pract. 2016 Nov;16(8):1064-1072. doi: 10.1111/papr.12407. Epub 2016 Feb 16. PMID 26878998
- [Background] Evans S, Seidman LC, Tsao JC, Lung KC, Zeltzer LK, Naliboff BD. Heart rate variability as a biomarker for autonomic nervous system response differences between children with chronic pain and healthy control children. J Pain Res. 2013 Jun 12;6:449-57. doi: 10.2147/JPR.S43849. Print 2013. PMID 23788839
- [Background] Sesay M, Robin G, Tauzin-Fin P, Sacko O, Gimbert E, Vignes JR, Liguoro D, Nouette-Gaulain K. Responses of heart rate variability to acute pain after minor spinal surgery: optimal thresholds and correlation with the numeric rating scale. J Neurosurg Anesthesiol. 2015 Apr;27(2):148-54. doi: 10.1097/ANA.0000000000000102. PMID 25105826
- [Background] Zeidan F, Vago DR. Mindfulness meditation-based pain relief: a mechanistic account. Ann N Y Acad Sci. 2016 Jun;1373(1):114-27. doi: 10.1111/nyas.13153. PMID 27398643
- [Background] Zeidan F, Adler-Neal AL, Wells RE, Stagnaro E, May LM, Eisenach JC, McHaffie JG, Coghill RC. Mindfulness-Meditation-Based Pain Relief Is Not Mediated by Endogenous Opioids. J Neurosci. 2016 Mar 16;36(11):3391-7. doi: 10.1523/JNEUROSCI.4328-15.2016. PMID 26985045
- [Background] Zeidan F, Emerson NM, Farris SR, Ray JN, Jung Y, McHaffie JG, Coghill RC. Mindfulness Meditation-Based Pain Relief Employs Different Neural Mechanisms Than Placebo and Sham Mindfulness Meditation-Induced Analgesia. J Neurosci. 2015 Nov 18;35(46):15307-25. doi: 10.1523/JNEUROSCI.2542-15.2015. PMID 26586819
- [Background] Brown ML, Rojas E, Gouda S. A Mind-Body Approach to Pediatric Pain Management. Children (Basel). 2017 Jun 20;4(6):50. doi: 10.3390/children4060050. PMID 28632194
- [Background] Dowsey MM, Castle DJ, Knowles SR, Monshat K, Salzberg MR, Choong PF. The effect of mindfulness training prior to total joint arthroplasty on post-operative pain and physical function: study protocol for a randomised controlled trial. Trials. 2014 Jun 5;15:208. doi: 10.1186/1745-6215-15-208. PMID 24899242
- [Background] Sanger KL, Dorjee D. Mindfulness training for adolescents: A neurodevelopmental perspective on investigating modifications in attention and emotion regulation using event-related brain potentials. Cogn Affect Behav Neurosci. 2015 Sep;15(3):696-711. doi: 10.3758/s13415-015-0354-7. PMID 25846954
- [Background] Shahidi S, Akbari H, Zargar F. Effectiveness of mindfulness-based stress reduction on emotion regulation and test anxiety in female high school students. J Educ Health Promot. 2017 Oct 4;6:87. doi: 10.4103/jehp.jehp_98_16. eCollection 2017. PMID 29114555
- [Background] Malboeuf-Hurtubise C, Lacourse E, Herba C, Taylor G, Amor LB. Mindfulness-based Intervention in Elementary School Students With Anxiety and Depression: A Series of n-of-1 Trials on Effects and Feasibility. J Evid Based Complementary Altern Med. 2017 Oct;22(4):856-869. doi: 10.1177/2156587217726682. Epub 2017 Aug 30. PMID 28853297
- [Background] Dariotis JK, Mirabal-Beltran R, Cluxton-Keller F, Gould LF, Greenberg MT, Mendelson T. A Qualitative Exploration of Implementation Factors in a School-Based Mindfulness and Yoga Program: Lessons Learned from Students and Teachers. Psychol Sch. 2017 Jan;54(1):53-69. doi: 10.1002/pits.21979. Epub 2016 Nov 28. PMID 28670007
- [Background] Gouda S, Luong MT, Schmidt S, Bauer J. Students and Teachers Benefit from Mindfulness-Based Stress Reduction in a School-Embedded Pilot Study. Front Psychol. 2016 Apr 26;7:590. doi: 10.3389/fpsyg.2016.00590. eCollection 2016. PMID 27199825
- [Background] Parker AE, Kupersmidt JB, Mathis ET, Scull TM, Sims C. The impact of mindfulness education on elementary school students: Evaluation of the Master Mind Program. Adv Sch Ment Health Promot. 2014;7(3):184-204. doi: 10.1080/1754730X.2014.916497. Epub 2014 May 19. PMID 27057208
- [Background] Holzel BK, Lazar SW, Gard T, Schuman-Olivier Z, Vago DR, Ott U. How Does Mindfulness Meditation Work? Proposing Mechanisms of Action From a Conceptual and Neural Perspective. Perspect Psychol Sci. 2011 Nov;6(6):537-59. doi: 10.1177/1745691611419671. PMID 26168376
- [Background] Dowman R. The role of the pain-evoked negative difference potential in dual-task response conflict. Eur J Pain. 2004 Dec;8(6):567-78. doi: 10.1016/j.ejpain.2004.02.001. PMID 15531225
- [Background] Pralong E, Pollo C, Bloch J, Villemure JG, Daniel RT, Tetreault MH, Debatisse D. Recording of ventral posterior lateral thalamus neuron response to contact heat evoked potential in patient with neurogenic pain. Neurosci Lett. 2004 Sep 9;367(3):332-5. doi: 10.1016/j.neulet.2004.06.024. PMID 15337260
- [Background] Dowman R. Pain-evoked anterior cingulate activity generating the negative difference potential may reflect response selection processes. Psychophysiology. 2002 May;39(3):369-79. doi: 10.1017/s0048577201393113. PMID 12212656
- [Background] Bhayee S, Tomaszewski P, Lee DH, Moffat G, Pino L, Moreno S, Farb NA. Attentional and affective consequences of technology supported mindfulness training: a randomised, active control, efficacy trial. BMC Psychol. 2016 Nov 29;4(1):60. doi: 10.1186/s40359-016-0168-6. PMID 27894358
- [Background] Karydis T, Aguiar F, Foster SL, Mershin A. Performance Characterization of Self-Calibrating Protocols for Wearable EEG Applications. Proceedings of the 8th ACM International Conference on PErvasive Technologies Related to Assistive Environments; 2015; Corfu, Greece: ACM, New York; 2015.
- [Background] Lee YH, Shiah YJ, Chen SC, Wang SF, Young MS, Lin CL. Improved emotional stability in experienced meditators with concentrative meditation based on electroencephalography and heart rate variability. J Altern Complement Med. 2015 Jan;21(1):31-9. doi: 10.1089/acm.2013.0465. Epub 2014 Oct 29. PMID 25354314
- [Background] Al-Fahoum AS, Al-Fraihat AA. Methods of EEG signal features extraction using linear analysis in frequency and time-frequency domains. ISRN Neurosci. 2014 Feb 13;2014:730218. doi: 10.1155/2014/730218. eCollection 2014. PMID 24967316
- [Background] Cotton S, Luberto CM, Bogenschutz LH, Pelley TJ, Dusek J. Integrative care therapies and pain in hospitalized children and adolescents: a retrospective database review. J Altern Complement Med. 2014 Feb;20(2):98-102. doi: 10.1089/acm.2013.0306. Epub 2013 Oct 31. PMID 24175871
- [Background] Chidambaran V, Ding L, Moore DL, Spruance K, Cudilo EM, Pilipenko V, Hossain M, Sturm P, Kashikar-Zuck S, Martin LJ, Sadhasivam S. Predicting the pain continuum after adolescent idiopathic scoliosis surgery: A prospective cohort study. Eur J Pain. 2017 Aug;21(7):1252-1265. doi: 10.1002/ejp.1025. Epub 2017 Mar 27. PMID 28346762
- [Background] Kimchi-Sarfaty C, Marple AH, Shinar S, Kimchi AM, Scavo D, Roma MI, Kim IW, Jones A, Arora M, Gribar J, Gurwitz D, Gottesman MM. Ethnicity-related polymorphisms and haplotypes in the human ABCB1 gene. Pharmacogenomics. 2007 Jan;8(1):29-39. doi: 10.2217/14622416.8.1.29. PMID 17187507
- [Background] Marshall-Gradisnik S, Johnston S, Chacko A, Nguyen T, Smith P, Staines D. Single nucleotide polymorphisms and genotypes of transient receptor potential ion channel and acetylcholine receptor genes from isolated B lymphocytes in myalgic encephalomyelitis/chronic fatigue syndrome patients. J Int Med Res. 2016 Dec;44(6):1381-1394. doi: 10.1177/0300060516671622. Epub 2016 Nov 11. PMID 27834303
- [Background] Owen GI, Richer JK, Tung L, Takimoto G, Horwitz KB. Progesterone regulates transcription of the p21(WAF1) cyclin- dependent kinase inhibitor gene through Sp1 and CBP/p300. J Biol Chem. 1998 Apr 24;273(17):10696-701. doi: 10.1074/jbc.273.17.10696. PMID 9553133
- [Background] Seo S, Grzenda A, Lomberk G, Ou XM, Cruciani RA, Urrutia R. Epigenetics: a promising paradigm for better understanding and managing pain. J Pain. 2013 Jun;14(6):549-57. doi: 10.1016/j.jpain.2013.01.772. Epub 2013 Apr 19. PMID 23602266
- [Background] Koch CM, Andrews RM, Flicek P, Dillon SC, Karaoz U, Clelland GK, Wilcox S, Beare DM, Fowler JC, Couttet P, James KD, Lefebvre GC, Bruce AW, Dovey OM, Ellis PD, Dhami P, Langford CF, Weng Z, Birney E, Carter NP, Vetrie D, Dunham I. The landscape of histone modifications across 1% of the human genome in five human cell lines. Genome Res. 2007 Jun;17(6):691-707. doi: 10.1101/gr.5704207. PMID 17567990
- [Background] Barski A, Cuddapah S, Cui K, Roh TY, Schones DE, Wang Z, Wei G, Chepelev I, Zhao K. High-resolution profiling of histone methylations in the human genome. Cell. 2007 May 18;129(4):823-37. doi: 10.1016/j.cell.2007.05.009. PMID 17512414
- [Background] Creyghton MP, Cheng AW, Welstead GG, Kooistra T, Carey BW, Steine EJ, Hanna J, Lodato MA, Frampton GM, Sharp PA, Boyer LA, Young RA, Jaenisch R. Histone H3K27ac separates active from poised enhancers and predicts developmental state. Proc Natl Acad Sci U S A. 2010 Dec 14;107(50):21931-6. doi: 10.1073/pnas.1016071107. Epub 2010 Nov 24. PMID 21106759
- [Background] Sadhasivam S, Chidambaran V, Ngamprasertwong P, Esslinger HR, Prows C, Zhang X, Martin LJ, McAuliffe J. Race and unequal burden of perioperative pain and opioid related adverse effects in children. Pediatrics. 2012 May;129(5):832-8. doi: 10.1542/peds.2011-2607. Epub 2012 Apr 23. PMID 22529273
- [Background] Sadhasivam S, Chidambaran V, Zhang X, Meller J, Esslinger H, Zhang K, Martin LJ, McAuliffe J. Opioid-induced respiratory depression: ABCB1 transporter pharmacogenetics. Pharmacogenomics J. 2015 Apr;15(2):119-26. doi: 10.1038/tpj.2014.56. Epub 2014 Oct 14. PMID 25311385
- [Background] Sadhasivam S, Chidambaran V. Pharmacogenomics of opioids and perioperative pain management. Pharmacogenomics. 2012 Nov;13(15):1719-40. doi: 10.2217/pgs.12.152. PMID 23171337
- [Background] Sadhasivam S, Krekels EH, Chidambaran V, Esslinger HR, Ngamprasertwong P, Zhang K, Fukuda T, Vinks AA. Morphine clearance in children: does race or genetics matter? J Opioid Manag. 2012 Jul-Aug;8(4):217-26. doi: 10.5055/jom.2012.0119. PMID 22941849
- [Background] Subramanyam R, Varughese A, Willging JP, Sadhasivam S. Future of pediatric tonsillectomy and perioperative outcomes. Int J Pediatr Otorhinolaryngol. 2013 Feb;77(2):194-9. doi: 10.1016/j.ijporl.2012.10.016. Epub 2012 Nov 16. PMID 23159321
- [Background] Fukuda T, Chidambaran V, Mizuno T, Venkatasubramanian R, Ngamprasertwong P, Olbrecht V, Esslinger HR, Vinks AA, Sadhasivam S. OCT1 genetic variants influence the pharmacokinetics of morphine in children. Pharmacogenomics. 2013 Jul;14(10):1141-51. doi: 10.2217/pgs.13.94. PMID 23859569
- [Background] Patino M, Sadhasivam S, Mahmoud M. Obstructive sleep apnoea in children: perioperative considerations. Br J Anaesth. 2013 Dec;111 Suppl 1:i83-95. doi: 10.1093/bja/aet371. PMID 24335402
- [Background] Prows CA, Zhang X, Huth MM, Zhang K, Saldana SN, Daraiseh NM, Esslinger HR, Freeman E, Greinwald JH, Martin LJ, Sadhasivam S. Codeine-related adverse drug reactions in children following tonsillectomy: a prospective study. Laryngoscope. 2014 May;124(5):1242-50. doi: 10.1002/lary.24455. Epub 2013 Nov 13. PMID 24122716
- [Background] Subramanyam R, Chidambaran V, Ding L, Myer CM 3rd, Sadhasivam S. Anesthesia- and opioids-related malpractice claims following tonsillectomy in USA: LexisNexis claims database 1984-2012. Paediatr Anaesth. 2014 Apr;24(4):412-20. doi: 10.1111/pan.12342. Epub 2014 Jan 13. PMID 24417679
- [Background] Crews KR, Gaedigk A, Dunnenberger HM, Leeder JS, Klein TE, Caudle KE, Haidar CE, Shen DD, Callaghan JT, Sadhasivam S, Prows CA, Kharasch ED, Skaar TC; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium guidelines for cytochrome P450 2D6 genotype and codeine therapy: 2014 update. Clin Pharmacol Ther. 2014 Apr;95(4):376-82. doi: 10.1038/clpt.2013.254. Epub 2014 Jan 23. PMID 24458010
- [Background] Sadhasivam S, Chidambaran V, Olbrecht VA, Esslinger HR, Zhang K, Zhang X, Martin LJ. Genetics of pain perception, COMT and postoperative pain management in children. Pharmacogenomics. 2014 Feb;15(3):277-84. doi: 10.2217/pgs.13.248. PMID 24533707
- [Background] Wang C, Sadhavisvam S, Krekels EH, Dahan A, Tibboel D, Danhof M, Vinks AA, Knibbe CA. Developmental changes in morphine clearance across the entire paediatric age range are best described by a bodyweight-dependent exponent model. Clin Drug Investig. 2013 Jul;33(7):523-34. doi: 10.1007/s40261-013-0097-6. PMID 23754691
- [Background] Venkatasubramanian R, Fukuda T, Niu J, Mizuno T, Chidambaran V, Vinks AA, Sadhasivam S. ABCC3 and OCT1 genotypes influence pharmacokinetics of morphine in children. Pharmacogenomics. 2014 Jul;15(10):1297-309. doi: 10.2217/pgs.14.99. PMID 25155932
- [Background] Chidambaran V, Mavi J, Esslinger H, Pilipenko V, Martin LJ, Zhang K, Sadhasivam S. Association of OPRM1 A118G variant with risk of morphine-induced respiratory depression following spine fusion in adolescents. Pharmacogenomics J. 2015 Jun;15(3):255-62. doi: 10.1038/tpj.2014.59. Epub 2014 Sep 30. PMID 25266679
- [Background] Biesiada J, Chidambaran V, Wagner M, Zhang X, Martin LJ, Meller J, Sadhasivam S. Genetic risk signatures of opioid-induced respiratory depression following pediatric tonsillectomy. Pharmacogenomics. 2014 Nov;15(14):1749-1762. doi: 10.2217/pgs.14.137. PMID 25493568
- [Background] Lotta T, Vidgren J, Tilgmann C, Ulmanen I, Melen K, Julkunen I, Taskinen J. Kinetics of human soluble and membrane-bound catechol O-methyltransferase: a revised mechanism and description of the thermolabile variant of the enzyme. Biochemistry. 1995 Apr 4;34(13):4202-10. doi: 10.1021/bi00013a008. PMID 7703232
- [Background] Caldas JC, Pais-Ribeiro JL, Carneiro SR. General anesthesia, surgery and hospitalization in children and their effects upon cognitive, academic, emotional and sociobehavioral development - a review. Paediatr Anaesth. 2004 Nov;14(11):910-5. doi: 10.1111/j.1460-9592.2004.01350.x. PMID 15500489
- [Background] McGraw T. Preparing children for the operating room: psychological issues. Can J Anaesth. 1994 Nov;41(11):1094-103. doi: 10.1007/BF03015661. PMID 7828259
- [Background] Devane WA, Hanus L, Breuer A, Pertwee RG, Stevenson LA, Griffin G, Gibson D, Mandelbaum A, Etinger A, Mechoulam R. Isolation and structure of a brain constituent that binds to the cannabinoid receptor. Science. 1992 Dec 18;258(5090):1946-9. doi: 10.1126/science.1470919.
- [Background] Van Sickle MD, Oland LD, Ho W, Hillard CJ, Mackie K, Davison JS, Sharkey KA. Cannabinoids inhibit emesis through CB1 receptors in the brainstem of the ferret. Gastroenterology. 2001 Oct;121(4):767-74. doi: 10.1053/gast.2001.28466. PMID 11606489
- [Background] Sipe JC, Chiang K, Gerber AL, Beutler E, Cravatt BF. A missense mutation in human fatty acid amide hydrolase associated with problem drug use. Proc Natl Acad Sci U S A. 2002 Jun 11;99(12):8394-9. doi: 10.1073/pnas.082235799. PMID 12060782
- [Background] Chiang KP, Gerber AL, Sipe JC, Cravatt BF. Reduced cellular expression and activity of the P129T mutant of human fatty acid amide hydrolase: evidence for a link between defects in the endocannabinoid system and problem drug use. Hum Mol Genet. 2004 Sep 15;13(18):2113-9. doi: 10.1093/hmg/ddh216. Epub 2004 Jul 14. PMID 15254019
- [Background] Lotsch J, Geisslinger G. Are mu-opioid receptor polymorphisms important for clinical opioid therapy? Trends Mol Med. 2005 Feb;11(2):82-9. doi: 10.1016/j.molmed.2004.12.006. PMID 15694871
- [Background] Bond C, LaForge KS, Tian M, Melia D, Zhang S, Borg L, Gong J, Schluger J, Strong JA, Leal SM, Tischfield JA, Kreek MJ, Yu L. Single-nucleotide polymorphism in the human mu opioid receptor gene alters beta-endorphin binding and activity: possible implications for opiate addiction. Proc Natl Acad Sci U S A. 1998 Aug 4;95(16):9608-13. doi: 10.1073/pnas.95.16.9608. PMID 9689128
- [Background] Romberg RR, Olofsen E, Bijl H, Taschner PE, Teppema LJ, Sarton EY, van Kleef JW, Dahan A. Polymorphism of mu-opioid receptor gene (OPRM1:c.118A>G) does not protect against opioid-induced respiratory depression despite reduced analgesic response. Anesthesiology. 2005 Mar;102(3):522-30. doi: 10.1097/00000542-200503000-00008. PMID 15731588
- [Background] Sia AT, Lim Y, Lim EC, Goh RW, Law HY, Landau R, Teo YY, Tan EC. A118G single nucleotide polymorphism of human mu-opioid receptor gene influences pain perception and patient-controlled intravenous morphine consumption after intrathecal morphine for postcesarean analgesia. Anesthesiology. 2008 Sep;109(3):520-6. doi: 10.1097/ALN.0b013e318182af21. PMID 18719451
- [Background] Sadhasivam S, Cohen LL, Szabova A, Varughese A, Kurth CD, Willging P, Wang Y, Nick TG, Gunter J. Real-time assessment of perioperative behaviors and prediction of perioperative outcomes. Anesth Analg. 2009 Mar;108(3):822-6. doi: 10.1213/ane.0b013e318195c115. PMID 19224789
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Bringuier S, Dadure C, Raux O, Dubois A, Picot MC, Capdevila X. The perioperative validity of the visual analog anxiety scale in children: a discriminant and useful instrument in routine clinical practice to optimize postoperative pain management. Anesth Analg. 2009 Sep;109(3):737-44. doi: 10.1213/ane.0b013e3181af00e4. PMID 19690240
- [Background] Chen E, Zeltzer LK, Craske MG, Katz ER. Alteration of memory in the reduction of children's distress during repeated aversive medical procedures. J Consult Clin Psychol. 1999 Aug;67(4):481-90. doi: 10.1037//0022-006x.67.4.481. PMID 10450618
- [Background] von Baeyer CL. Numerical rating scale for self-report of pain intensity in children and adolescents: recent progress and further questions. Eur J Pain. 2009 Nov;13(10):1005-7. doi: 10.1016/j.ejpain.2009.08.006. Epub 2009 Sep 17. No abstract available. PMID 19766028
- [Background] von Baeyer CL, Spagrud LJ, McCormick JC, Choo E, Neville K, Connelly MA. Three new datasets supporting use of the Numerical Rating Scale (NRS-11) for children's self-reports of pain intensity. Pain. 2009 Jun;143(3):223-227. doi: 10.1016/j.pain.2009.03.002. Epub 2009 Apr 8. PMID 19359097
- [Background] Bulloch B, Tenenbein M. Validation of 2 pain scales for use in the pediatric emergency department. Pediatrics. 2002 Sep;110(3):e33. doi: 10.1542/peds.110.3.e33. PMID 12205283
- [Background] Voepel-Lewis T, Marinkovic A, Kostrzewa A, Tait AR, Malviya S. The prevalence of and risk factors for adverse events in children receiving patient-controlled analgesia by proxy or patient-controlled analgesia after surgery. Anesth Analg. 2008 Jul;107(1):70-5. doi: 10.1213/ane.0b013e318172fa9e. PMID 18635469
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] Ramsay MA. Anesthesia and pain management at Baylor University Medical Center. Proc (Bayl Univ Med Cent). 2000 Apr;13(2):151-65. doi: 10.1080/08998280.2000.11927660. No abstract available. PMID 16389370
- [Background] Aubrun F, Monsel S, Langeron O, Coriat P, Riou B. Postoperative titration of intravenous morphine. Eur J Anaesthesiol. 2001 Mar;18(3):159-65. doi: 10.1046/j.0265-0215.2000.00796.x. PMID 11298174
- [Background] Paqueron X, Lumbroso A, Mergoni P, Aubrun F, Langeron O, Coriat P, Riou B. Is morphine-induced sedation synonymous with analgesia during intravenous morphine titration? Br J Anaesth. 2002 Nov;89(5):697-701. PMID 12393765
- [Background] Silverman WK, Goedhart AW, Barrett P, Turner C. The facets of anxiety sensitivity represented in the childhood anxiety sensitivity index: confirmatory analyses of factor models from past studies. J Abnorm Psychol. 2003 Aug;112(3):364-74. doi: 10.1037/0021-843x.112.3.364. PMID 12943015
- [Background] Walker LS, Greene JW. The functional disability inventory: measuring a neglected dimension of child health status. J Pediatr Psychol. 1991 Feb;16(1):39-58. doi: 10.1093/jpepsy/16.1.39. PMID 1826329
- [Background] Kashikar-Zuck S, Vaught MH, Goldschneider KR, Graham TB, Miller JC. Depression, coping, and functional disability in juvenile primary fibromyalgia syndrome. J Pain. 2002 Oct;3(5):412-9. doi: 10.1054/jpai.2002.126786. PMID 14622745
- [Background] Kashikar-Zuck S, Flowers SR, Claar RL, Guite JW, Logan DE, Lynch-Jordan AM, Palermo TM, Wilson AC. Clinical utility and validity of the Functional Disability Inventory among a multicenter sample of youth with chronic pain. Pain. 2011 Jul;152(7):1600-1607. doi: 10.1016/j.pain.2011.02.050. Epub 2011 Mar 31. PMID 21458162
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849
- [Background] Freynhagen R, Tolle TR, Gockel U, Baron R. The painDETECT project - far more than a screening tool on neuropathic pain. Curr Med Res Opin. 2016 Jun;32(6):1033-57. doi: 10.1185/03007995.2016.1157460. Epub 2016 Mar 11. PMID 26907456
- [Background] Desai AD, Zhou C, Stanford S, Haaland W, Varni JW, Mangione-Smith RM. Validity and responsiveness of the pediatric quality of life inventory (PedsQL) 4.0 generic core scales in the pediatric inpatient setting. JAMA Pediatr. 2014 Dec;168(12):1114-21. doi: 10.1001/jamapediatrics.2014.1600. PMID 25347549
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Kashikar-Zuck S, Goldschneider KR, Powers SW, Vaught MH, Hershey AD. Depression and functional disability in chronic pediatric pain. Clin J Pain. 2001 Dec;17(4):341-9. doi: 10.1097/00002508-200112000-00009. PMID 11783815
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Irwin DE, Stucky B, Langer MM, Thissen D, Dewitt EM, Lai JS, Varni JW, Yeatts K, DeWalt DA. An item response analysis of the pediatric PROMIS anxiety and depressive symptoms scales. Qual Life Res. 2010 May;19(4):595-607. doi: 10.1007/s11136-010-9619-3. Epub 2010 Mar 7. PMID 20213516
- [Background] Reid GJ, Gilbert CA, McGrath PJ. The Pain Coping Questionnaire: preliminary validation. Pain. 1998 May;76(1-2):83-96. doi: 10.1016/s0304-3959(98)00029-3. PMID 9696461
- [Background] Cunningham NR, Kashikar-Zuck S, Mara C, Goldschneider KR, Revicki DA, Dampier C, Sherry DD, Crosby L, Carle A, Cook KF, Morgan EM. Development and validation of the self-reported PROMIS pediatric pain behavior item bank and short form scale. Pain. 2017 Jul;158(7):1323-1331. doi: 10.1097/j.pain.0000000000000914. PMID 28394851
- [Background] Amtmann D, Cook KF, Jensen MP, Chen WH, Choi S, Revicki D, Cella D, Rothrock N, Keefe F, Callahan L, Lai JS. Development of a PROMIS item bank to measure pain interference. Pain. 2010 Jul;150(1):173-182. doi: 10.1016/j.pain.2010.04.025. PMID 20554116
- [Background] Lai JS, Stucky BD, Thissen D, Varni JW, DeWitt EM, Irwin DE, Yeatts KB, DeWalt DA. Development and psychometric properties of the PROMIS((R)) pediatric fatigue item banks. Qual Life Res. 2013 Nov;22(9):2417-27. doi: 10.1007/s11136-013-0357-1. Epub 2013 Feb 2. PMID 23378106
- [Background] Dewalt DA, Thissen D, Stucky BD, Langer MM, Morgan Dewitt E, Irwin DE, Lai JS, Yeatts KB, Gross HE, Taylor O, Varni JW. PROMIS Pediatric Peer Relationships Scale: development of a peer relationships item bank as part of social health measurement. Health Psychol. 2013 Oct;32(10):1093-103. doi: 10.1037/a0032670. Epub 2013 Jun 17. PMID 23772887
- [Background] Carver CS, & White, TL. Behavioral inhibition, behavioral activation, and affective responses to impending reward and punishment: The BIS/BAS scales. Journal of Personality and Social Psychology 1994; 67(2): 319-333.
- [Background] Webster LR, Webster RM. Predicting aberrant behaviors in opioid-treated patients: preliminary validation of the Opioid Risk Tool. Pain Med. 2005 Nov-Dec;6(6):432-42. doi: 10.1111/j.1526-4637.2005.00072.x. PMID 16336480
- [Background] Knight JR, Sherritt L, Shrier LA, Harris SK, Chang G. Validity of the CRAFFT substance abuse screening test among adolescent clinic patients. Arch Pediatr Adolesc Med. 2002 Jun;156(6):607-14. doi: 10.1001/archpedi.156.6.607. PMID 12038895
- [Background] Greco LA, Baer RA, Smith GT. Assessing mindfulness in children and adolescents: development and validation of the Child and Adolescent Mindfulness Measure (CAMM). Psychol Assess. 2011 Sep;23(3):606-14. doi: 10.1037/a0022819. PMID 21480722
- [Background] Crombez G, Bijttebier P, Eccleston C, Mascagni T, Mertens G, Goubert L, Verstraeten K. The child version of the pain catastrophizing scale (PCS-C): a preliminary validation. Pain. 2003 Aug;104(3):639-646. doi: 10.1016/S0304-3959(03)00121-0. PMID 12927636
- [Background] Kashikar-Zuck S, Lynch AM, Slater S, Graham TB, Swain NF, Noll RB. Family factors, emotional functioning, and functional impairment in juvenile fibromyalgia syndrome. Arthritis Rheum. 2008 Oct 15;59(10):1392-8. doi: 10.1002/art.24099. PMID 18821640
- [Background] Van Slyke DA, Walker LS. Mothers' responses to children's pain. Clin J Pain. 2006 May;22(4):387-91. doi: 10.1097/01.ajp.0000205257.80044.01. PMID 16691093
- [Background] Cunningham NR, Lynch-Jordan A, Barnett K, Peugh J, Sil S, Goldschneider K, Kashikar-Zuck S. Child pain catastrophizing mediates the relation between parent responses to pain and disability in youth with functional abdominal pain. J Pediatr Gastroenterol Nutr. 2014 Dec;59(6):732-8. doi: 10.1097/MPG.0000000000000529. PMID 25121521
- [Background] Law EF, Dufton L, Palermo TM. Daytime and nighttime sleep patterns in adolescents with and without chronic pain. Health Psychol. 2012 Nov;31(6):830-3. doi: 10.1037/a0026485. Epub 2011 Dec 12. PMID 22149126
- [Background] van de Water AT, Eadie J, Hurley DA. Investigation of sleep disturbance in chronic low back pain: an age- and gender-matched case-control study over a 7-night period. Man Ther. 2011 Dec;16(6):550-6. doi: 10.1016/j.math.2011.05.004. Epub 2011 Jun 8. PMID 21652257
- [Background] O'Brien EM, Waxenberg LB, Atchison JW, Gremillion HA, Staud RM, McCrae CS, Robinson ME. Intraindividual variability in daily sleep and pain ratings among chronic pain patients: bidirectional association and the role of negative mood. Clin J Pain. 2011 Jun;27(5):425-33. doi: 10.1097/AJP.0b013e318208c8e4. PMID 21415723
- [Background] Zeidan F, Johnson SK, Diamond BJ, David Z, Goolkasian P. Mindfulness meditation improves cognition: evidence of brief mental training. Conscious Cogn. 2010 Jun;19(2):597-605. doi: 10.1016/j.concog.2010.03.014. Epub 2010 Apr 3. PMID 20363650
- [Background] Zeidan F, Gordon NS, Merchant J, Goolkasian P. The effects of brief mindfulness meditation training on experimentally induced pain. J Pain. 2010 Mar;11(3):199-209. doi: 10.1016/j.jpain.2009.07.015. Epub 2009 Oct 22. PMID 19853530
- [Background] Shapiro DH Jr. Adverse effects of meditation: a preliminary investigation of long-term meditators. Int J Psychosom. 1992;39(1-4):62-7. PMID 1428622
- [Background] Landman Z, Oswald T, Sanders J, Diab M; Spinal Deformity Study Group. Prevalence and predictors of pain in surgical treatment of adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2011 May 1;36(10):825-9. doi: 10.1097/BRS.0b013e3181de8c2b. PMID 21192302
- [Background] Price AL, Patterson NJ, Plenge RM, Weinblatt ME, Shadick NA, Reich D. Principal components analysis corrects for stratification in genome-wide association studies. Nat Genet. 2006 Aug;38(8):904-9. doi: 10.1038/ng1847. Epub 2006 Jul 23. PMID 16862161
- [Background] Bursac Z, Gauss CH, Williams DK, Hosmer DW. Purposeful selection of variables in logistic regression. Source Code Biol Med. 2008 Dec 16;3:17. doi: 10.1186/1751-0473-3-17. PMID 19087314
- [Background] Chen H, Wang C, Conomos MP, Stilp AM, Li Z, Sofer T, Szpiro AA, Chen W, Brehm JM, Celedon JC, Redline S, Papanicolaou GJ, Thornton TA, Laurie CC, Rice K, Lin X. Control for Population Structure and Relatedness for Binary Traits in Genetic Association Studies via Logistic Mixed Models. Am J Hum Genet. 2016 Apr 7;98(4):653-66. doi: 10.1016/j.ajhg.2016.02.012. Epub 2016 Mar 24. PMID 27018471
- [Background] Moore JH. Analysis of gene-gene interactions. Curr Protoc Hum Genet. 2004 Feb;Chapter 1:Unit 1.14. doi: 10.1002/0471142905.hg0114s39. PMID 18428353
- [Background] Sun G, Kaushal R, Pal P, Wolujewicz M, Smelser D, Cheng H, Lu M, Chakraborty R, Jin L, Deka R. Whole-genome amplification: relative efficiencies of the current methods. Leg Med (Tokyo). 2005 Oct;7(5):279-86. doi: 10.1016/j.legalmed.2005.05.001. PMID 15990351
- [Background] Chizarifard A. SEM Analysis of Epigenetic Data. Uppsala: Uppsala University; 2014.
- [Background] Du P, Zhang X, Huang CC, Jafari N, Kibbe WA, Hou L, Lin SM. Comparison of Beta-value and M-value methods for quantifying methylation levels by microarray analysis. BMC Bioinformatics. 2010 Nov 30;11:587. doi: 10.1186/1471-2105-11-587. PMID 21118553
- [Background] Maurano MT, Humbert R, Rynes E, Thurman RE, Haugen E, Wang H, Reynolds AP, Sandstrom R, Qu H, Brody J, Shafer A, Neri F, Lee K, Kutyavin T, Stehling-Sun S, Johnson AK, Canfield TK, Giste E, Diegel M, Bates D, Hansen RS, Neph S, Sabo PJ, Heimfeld S, Raubitschek A, Ziegler S, Cotsapas C, Sotoodehnia N, Glass I, Sunyaev SR, Kaul R, Stamatoyannopoulos JA. Systematic localization of common disease-associated variation in regulatory DNA. Science. 2012 Sep 7;337(6099):1190-5. doi: 10.1126/science.1222794. Epub 2012 Sep 5. PMID 22955828
- [Background] Hindorff LA, Sethupathy P, Junkins HA, Ramos EM, Mehta JP, Collins FS, Manolio TA. Potential etiologic and functional implications of genome-wide association loci for human diseases and traits. Proc Natl Acad Sci U S A. 2009 Jun 9;106(23):9362-7. doi: 10.1073/pnas.0903103106. Epub 2009 May 27. PMID 19474294
- [Background] ENCODE Project Consortium. An integrated encyclopedia of DNA elements in the human genome. Nature. 2012 Sep 6;489(7414):57-74. doi: 10.1038/nature11247. PMID 22955616
- [Background] Bernstein BE, Stamatoyannopoulos JA, Costello JF, Ren B, Milosavljevic A, Meissner A, Kellis M, Marra MA, Beaudet AL, Ecker JR, Farnham PJ, Hirst M, Lander ES, Mikkelsen TS, Thomson JA. The NIH Roadmap Epigenomics Mapping Consortium. Nat Biotechnol. 2010 Oct;28(10):1045-8. doi: 10.1038/nbt1010-1045. PMID 20944595
- [Background] Liu T, Ortiz JA, Taing L, Meyer CA, Lee B, Zhang Y, Shin H, Wong SS, Ma J, Lei Y, Pape UJ, Poidinger M, Chen Y, Yeung K, Brown M, Turpaz Y, Liu XS. Cistrome: an integrative platform for transcriptional regulation studies. Genome Biol. 2011 Aug 22;12(8):R83. doi: 10.1186/gb-2011-12-8-r83. PMID 21859476
- [Background] Griffon A, Barbier Q, Dalino J, van Helden J, Spicuglia S, Ballester B. Integrative analysis of public ChIP-seq experiments reveals a complex multi-cell regulatory landscape. Nucleic Acids Res. 2015 Feb 27;43(4):e27. doi: 10.1093/nar/gku1280. Epub 2014 Dec 3. PMID 25477382
- [Background] Whitlock MC. Combining probability from independent tests: the weighted Z-method is superior to Fisher's approach. J Evol Biol. 2005 Sep;18(5):1368-73. doi: 10.1111/j.1420-9101.2005.00917.x. PMID 16135132
- [Background] Krigolson OE, Williams CC, Norton A, Hassall CD, Colino FL. Choosing MUSE: Validation of a Low-Cost, Portable EEG System for ERP Research. Front Neurosci. 2017 Mar 10;11:109. doi: 10.3389/fnins.2017.00109. eCollection 2017. PMID 28344546
- [Background] Hall M, Frank E, Holmes G, Pfahringer B, Reutemann P, Witten IH. The WEKA data mining software: an update. ACM SIGKDD Explorations Newsletter 2009; 11(1): 10-8.